CLINICAL TRIAL: NCT04103138
Title: EEG Monitoring Under Anaesthesia in Children: Towards Personalized Anaesthesia Care
Acronym: EEGPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CIRB 2019/2235
Record Dates: First submitted 2019-08-25; First posted 2019-09-25 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2019-07

CONDITIONS: Depth of Anaesthesia; EEG; Anesthesia Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject and the outcome assessor analysing the EEG subsequently will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-Guided Anaesthesia (Experimental): Patients will have Sedline EEG sensor placed and anaesthesia guided by the EEG characteristics, patient state index (PSI) and suppression ratio (SR), in addition to routine clinical parameters.
  Interventions: Device: Sedline EEG sensor placement; Device: Sedline EEG monitoring
- Routine Care (Active Comparator): Patients will have Sedline EEG sensor placed but the monitor is concealed so the clinician is blinded to the EEG response. Anaesthesia is guided by routine clinical parameters.
  Interventions: Device: Sedline EEG sensor placement

INTERVENTIONS:
Device: Sedline EEG sensor placement — Patients will have Sedline EEG sensor placed before or immediately after induction.
Device: Sedline EEG monitoring — Anaesthesia depth will be guided by EEG characteristics in addition to routine clinical parameters
  Arms: EEG-Guided Anaesthesia

SUMMARY:
Electroencephalographic recordings (EEG) present an opportunity to monitor changes in human brain electrical activity during changing states of consciousness during general anesthesia.

The investigators aim to determine if EEG-guided anaesthesia using the Masimo Sedline Root monitor will result in different anaesthetic requirements, different anaesthetic depth, and emergence characteristics in children under 16 years of age.

200 children under 16 years undergoing routine general anaesthesia under sevoflurane will be randomized to either EEG monitoring or routine care. We will compare the anaesthetic requirements, the patient state index, number of episodes of burst suppression and the incidence and severity of emergence delrium between the two groups.

DETAILED DESCRIPTION:
Electroencephalographic recordings (EEG) present an opportunity to monitor changes in human brain electrical activity during changing states of consciousness during general anesthesia.

At present, monitoring of the brain under anaesthesia is not routinely employed. Since every patient is different and the way their brain response to anaesthetic drugs is different, it is important to adjust the patients' anaesthetic depth according to their brains' response, rather than only relying on routine cardiorespiratory parameters. This is important particularly for children, whose physiological responses and electroencephalographic recordings (EEG) differ from that of adults.

200 children under 16 years undergoing routine sevoflurane general anaesthesia will be randomized to either EEG-guided anaesthesia or routine care. The investigators will compare the anaesthetic requirements, the patient state index, number of episodes of burst suppression and the incidence and severity of emergence delrium between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 1-16 years old scheduled to undergo general sevoflurane anaesthesia for surgeries or procedures anticipated to last at between 30 minutes to 4 hours.

Exclusion Criteria:

* Patients with neurological diseases including seizure disorders
* Patients with developmental delay or genetic syndromes
* Patients with craniofacial deformities where it is not possible to place the EEG sensors
* Patients with severe eczema or skin allergy or atopy.
* Patients who are having craniofacial surgery where it is not possible to place the EEG sensors
* Patients whose foreheads are too small to accommodate the EEG sensors.
* Patients who require sedative premedications.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
End tidal sevoflurane concentration at induction | 6 hours: within the intraoperative period
  Average sevoflurane concentration (MAC) required during induction
End tidal sevoflurane concentration for maintenance | 6 hours: within the intraoperative period
  Average sevoflurane concentration (MAC) required during maintenance

SECONDARY OUTCOMES:
Emergence delirium incidence | Within 3 hours: Postoperative in PACU
  Incidence of emergence delirium as measured by the PAED scale
Emergence delirium severity | Within 3 hours: Postoperative in PACU
  Severity of emergence delirium as measured by the PAED scale
Post-operative behaviour | Within 2 weeks after surgery
  Post-operative maladaptive behaviour
Burst Suppression Incidence | 6 hours: within the intraoperative period
  Incidence of burst suppression
Burst Suppression Duration | 6 hours: within the intraoperative period
  Duration of burst suppression
Burst suppression probability | During maintenance of anaesthesia (up to 4 hours)
  Burst suppression probability during maintenance, summarized by the mean over the maintenance period
PSI | 6 hours: within the intraoperative period
  Patient state index during maintenance of anaesthesia

OTHER OUTCOMES:
Mean peak alpha frequency | During maintenance of anaesthesia (up to 4 hours)
  Mean peak alpha frequency during maintenance, computed in units of Hz by first searching for the frequency in the alpha band (8 to 12 Hz) that has maximum power in the spectrum, followed by computing the mean over the anesthetic maintenance period, which begins at the start of surgery and ends at the conclusion of the surgical procedure;
Mean peak alpha power | During maintenance of anaesthesia (up to 4 hours)
  Mean peak alpha power during maintenance, computed by calculating the mean power in the alpha band (8 to 12 Hz) in units of decibels (dB) during the anesthetic maintenance period which begins at the start of surgery and ends at the end of the surgical procedure;
Mean peak slow oscillation frequency | During maintenance of anaesthesia (up to 4 hours)
  Mean peak slow oscillation frequency during maintenance, computed in units of Hz by first searching for the frequency in the slowband (0.1-1 Hz) that has maximum power in the spectrum, followed by computing the mean over the anesthetic maintenance period, which begins at the start of surgery and ends at the conclusion of the surgical procedure;
Mean peak Slow oscillation power | During maintenance of anaesthesia (up to 4 hours)
  Mean peak Slow oscillation power during maintenance, computed by calculating the mean power in the slow band (0.1-1Hz) in units of decibels (dB) during the anesthetic maintenance period which begins at the start of surgery and ends at the end of the surgical procedure.
Variation in peak alpha frequency | During maintenance of anaesthesia (up to 4 hours)
  Variation in peak alpha frequency over time during maintenance, computed as the standard deviation of the mean peak alpha frequency, in units of Hz, during the anesthetic maintenance period which begins at the start of surgery and ends at the end of the surgical procedure.
Variation in peak alpha power | During maintenance of anaesthesia (up to 4 hours)
  Variation in peak alpha power over time during maintenance for each patient; computed as the standard deviation of the mean peak alpha power, in units of decibels, during the anesthetic maintenance period which begins at the start of surgery and ends at the end of the surgical procedure.
Phase amplitude modulation depth | During maintenance of anaesthesia (up to 4 hours)
  Phase amplitude modulation depth: The depth of phase amplitude modulation, as defined in Soulat, et al.., 2019, is a dimensionless number between 0 and 1 that describes the extent to which the amplitude of a higher frequency (alpha) oscillation is modulated by a lower frequency (slow) oscillation
  Soulat, H., Stephen, E. P., Beck, A. M., & Purdon, P. L. (2019). State Space Methods for Phase Amplitude Coupling Analysis [Preprint]. Neuroscience. https://doi.org/10.1101/772145
Phase amplitude modulation phase | During maintenance of anaesthesia (up to 4 hours)
  Phase amplitude modulation phase: The modulation phase, as defined in Soulat, et al.., 2019, is the phase, represented as an angle in units of degrees, that describes the lower frequency (slow) phase at which the amplitude of a higher frequency (alpha) oscillation is maximized.
  Soulat, H., Stephen, E. P., Beck, A. M., & Purdon, P. L. (2019). State Space Methods for Phase Amplitude Coupling Analysis [Preprint]. Neuroscience. https://doi.org/10.1101/772145

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No